CLINICAL TRIAL: NCT01564134
Title: Effect of Dose of Hepatitis B Vaccines in Non/Low-response Populations
Brief Title: Dose of Hepatitis B Vaccines in Non/Low-response Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wu Jiang (Other Government)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Sponsor-Investigator, Wu Jiang, Department of Immunization & Prevention, Centers for Disease Control and Prevention, China
Organization: Centers for Disease Control and Prevention, China (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BJCDCWJ201102
Record Dates: First submitted 2012-03-23; First posted 2012-03-27 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Vaccination; Complications, Reaction, Serum
Keywords: response vaccination
MeSH Terms: interventions — Hepatitis B Vaccines; gamma-hydroxy-gamma-ethyl-gamma-phenylbutyramide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- HepB 5ug (Experimental): receive the vaccine with 5ug HBsAg
  Interventions: Biological: hepatitis B vaccine
- HepB 10ug (Experimental): receive the vaccine with 10ug HBsAg
  Interventions: Biological: hepatitis B vaccine
- HepB 20ug (Experimental): receive the vaccine with 20ug HBsAg
  Interventions: Biological: hepatitis B vaccine
- HepB 60ug (Experimental): receive the vaccine with 60ug HBsAg
  Interventions: Biological: hepatitis B vaccine

INTERVENTIONS:
Biological: hepatitis B vaccine — hepatitis B vaccine with 5ug,10ug,20ug,60ug HBsAg
  Other Names: HepB 10ug: Hansenula Polymorpha Yeast; HepB 60ug: Saccharomyces cerevisiae

SUMMARY:
An interventional study will be performed in subjects aged 1-65 years old to evaluate effects of different doses of hepatitis B vaccines in low or non-response population.

DETAILED DESCRIPTION:
A randomized clinical study will be conducted to evaluate effects of different doses of hepatitis B vaccines in low or non-response population in China. 650 low or non-response subjects after hepatitis B vaccination will be enrolled under the premise of informed consent. 200 subjects aged 1-17 years will be divided into 3 groups and 450 subjects aged 18-65years will be divided into 4 groups. Group 1/2/3 will receive 3 doses of vaccine on day 0,30 and 180, with 5ug/10ug/20ug HBs-Ag respectively. Group 4 will receive 1 dose of vaccine with 60ug HBs-Ag, low or nonresponse subjects of which will receive the second dose by an interval of at least 28 days. All vaccinations will be done by specific study personnel, who do not take part in the assessment of safety or immunogenicity. Adverse events will be recorded after vaccination and blood samples were collected at day 30 after each vaccination for antibody detection.

The clinical program approved by the ethics committee will be performed by the researchers independently. Inspectors designated by the sponsor will take meticulous on-site audits to ensure the safety specifications during the whole process of research.

ELIGIBILITY:
Inclusion Criteria:

* aged 1-65 years old
* male or non-pregnant female volunteers
* provide written informed consents before joining the trial
* clinically healthy as determined by: medical history inquiring and physical examination
* negative for HBsAg,HBsAb,HBcAb,HBeAg,HBeAb within the past 1 year

Exclusion Criteria:

* No history of hepatitis B vaccine
* receipt of immunoglobulin within the past 1 month
* allergic to any ingredient of vaccine
* history of serious side effects, such as allergies, hives, breathing difficulties, angioedema or abdominal pain
* severe acute and chronic diseases
* autoimmune disease or immune deficiency
* axillary temperature > 37.0 ℃ over the time of vaccination

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 537 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Seroconversion rates of different doses of vaccines the levels of HBs-Ab after vaccination | day 30 after each vaccination
  describe the levels of HBs-Ab after each vaccination and compare the percentages of adverse events in all groups

CONTACTS AND LOCATIONS:
Overall Officials: jiang wu, Bachelor, Principal Investigator — Beijing Centers for Disease Control and Prevention
Locations (2):
- China (2):
  - Xicheng Centers For Disease Prevention & Control, Xicheng District, Beijing Municipality
  - Chifeng Centers For Disease Prevention & Control, Chifeng, Inner Mongolia